CLINICAL TRIAL: NCT01077999
Title: Chemoradiation Combined With Panitumumab Followed by Surgery for Patients With Operable Esophageal Cancer
Brief Title: Chemoradiation and Panitumumab for Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.W. Wilmink, Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCmedon08/381
Record Dates: First submitted 2010-02-25; First posted 2010-03-02 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Squamous Cell Carcinoma; Adenocarcinoma; Esophageal Cancer; Gastro-esophageal Junction Cancer
Keywords: chemoradiation; panitumumab; esophageal cancer; Resectable squamous cell carcinoma, adenocarcinoma or undifferentiated carcinoma of the intrathoracic esophagus or gastro esophageal junction
MeSH Terms: conditions — Carcinoma, Squamous Cell; Adenocarcinoma; Esophageal Neoplasms | interventions — Carboplatin; Paclitaxel; Panitumumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin + paclitaxel + radiotherapy (Active Comparator): Carboplatin AUC = 2, Paclitaxel 50 mg/m2 (both weekly) , a total dose of 41.4 Gy will be given in 23 fractions of 1.8 Gy.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: radiotherapy
- Carboplatin+ paclitaxel+ panitumumab+ radiotherapy (Experimental): Carboplatin AUC = 2, Paclitaxel 50 mg/m2 (both weekly) , a total dose of 41.4 Gy will be given in 23 fractions of 1.8 Gy. Panitumumab panitumumab: 6mg/kg in weeks 1-3-5.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: panitumumab; Radiation: radiotherapy

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC = 2 , weekly.
Drug: Paclitaxel — Paclitaxel 50 mg/m2, weekly
Drug: panitumumab — panitumumab: 6mg/kg in weeks 1-3-5.
  Other Names: vectibix
  Arms: Carboplatin+ paclitaxel+ panitumumab+ radiotherapy
Radiation: radiotherapy — A total dose of 41.4 Gy will be given in 23 fractions of 1.8 Gy.

SUMMARY:
A consistent finding in many studies in patients with operable esophageal and gastro-esophageal junction (GEJ) cancer is that response to preoperative therapy, particularly the absence of residual disease in the surgical specimen, is an indicator of better disease-free and overall survival. Therefore in the investigators trial the investigators will evaluate the pathologic response of panitumumab in combination with neoadjuvant chemoradiation as first line treatment of operable adenocarcinomas, undifferentiated or squamous cell carcinomas of the esophagus.

DETAILED DESCRIPTION:
This is a Phase II, non-randomized trial. Eligible subjects will be treated with panitumumab plus carboplatin, paclitaxel and radiotherapy followed by surgical resection of the esophagus.

Panitumumab administration schedule: Panitumumab will be administered as a 60-minute ± 15 minutes IV infusion, prior to administration of chemotherapy at a dose of 6 mg/kg on day 1, 15 and 29. If the first infusion is well tolerated (without any serious infusion related reactions) all subsequent infusions may be administered over 30 minutes ± 10 minutes.

Chemotherapy regimen: Paclitaxel 50 mg/m2 and Carboplatin AUC = 2 will be given by intravenous infusion on days 1, 8, 15, 22 and 29. Both drugs will be infused over one hour.

Radiotherapy treatment: A total dose of 41.4 Gy will be given in 23 fractions of 1.8 Gy, 5 fractions per week, starting the first day of the first cycle of chemotherapy. All patients will be radiated by external beam radiation, using 3-D conformal radiation technique.

Surgery: Surgery will be performed preferably within 6 weeks after the completion of the chemoradiation and panitumumab. For carcinomas distal of the tracheal bifurcation but proximal to the gastro-esophageal junction, a transthoracic approach is preferred. For distal tumors involving the gastro-esophageal junction a transhiatal esophageal resection is preferred. A wide local excision including the N1 lymph nodes is carried out in both techniques including a standard excision of the lymph nodes around the coeliac axis. The continuity of the digestive tract will be restored by a gastric tube reconstruction or colonic interposition procedure with an anastomosis in the neck.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma, adenocarcinoma or undifferentiated carcinoma of the intrathoracic esophagus or gastro esophageal junction
* Surgical resectable (T2-3, N0-1, M0), as determined by Endoscopic Ultra Sound (EUS) and CT scan of neck, thorax and abdomen.
* T1N1 tumors are eligible, T1N0 tumors and in situ carcinoma are not eligible
* Tumor length longitudinal ≤ 10 cm and radial ≤ 5 cm
* If tumor extends below the gastroesophageal (GE) junction into the proximal stomach, the bulk of the tumor must involve the esophagus or GE junction. The tumor must not extend more than 2 cm into the stomach. Gastric cancers with minor involvement of the GE junction or distal esophagus are not eligible
* No invasion of the tracheobronchial tree or presence of tracheoesophageal fistula
* Non pregnant, non-lactating female patients, not planning to become pregnant within 6 months after the end of treatment.
* Age ≥ 18 and ≤ 75
* ECOG performance status 0 or 1
* Adequate hematological, renal, hepatic and pulmonary functions
* Written, voluntary informed consent
* Patients must be accessible to follow up and management in the treatment center

Exclusion Criteria:

* Past or current history of malignancy other than entry diagnosis except for non-melanomatous skin cancer, or curatively treated in situ carcinoma of the cervix, or malignancy more than 5 years prior to enrollment
* Pregnancy (positive serum pregnancy test) and lactation
* Patient (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment
* Previous chemotherapy, radiotherapy, treatment with an anti-EGFR antibody or with small molecule EGFR inhibitors
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before randomization
* Pulmonary fibrosis
* Pre-existing motor or sensory neurotoxicity greater than WHO grade 1
* Active infection or other serious underlying medical condition which would impair the ability of the patient to receive the planned treatment, including prior allergic reactions to drugs containing Cremophor, such as teniposide or cyclosporine.
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent
* Inadequate caloric- and/or fluid intake
* Weight loss > 15%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Percentage of pathologic complete responses | 6 weeks after the completion of the chemoradiation

SECONDARY OUTCOMES:
R0 resection rate | the pathologist will determine the resection rate
Progression free survival | Every 3 months during the first 2 years after surgery, and every 6 months thereafter.
Toxicity profile | Weekly during chemoradiation. After surgery: every 3 months during the first 2 years after surgery, and every 6 months thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Wilmink, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands